CLINICAL TRIAL: NCT01740947
Title: Perioperative Selective Decontamination of the Digestive Tract (SDD) in Elective Colorectal Cancer Patients: a Multicenter Randomized Clinical Trial
Brief Title: Does Administration of Antibiotics in Patients Undergoing Surgery for Colorectal Cancer Result in Less Complications and Better Prognosis?
Acronym: SELECT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Superiority was no longer attainable
Sponsor: H. Jaap Bonjer, PhD (Other)
Collaborators: Dutch Digestive Diseases Foundation (Other)
Responsible Party: Sponsor-Investigator, H. Jaap Bonjer, PhD, Professor of Surgery, Amsterdam UMC, location VUmc
Organization: Amsterdam UMC, location VUmc (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011-002211-28
Record Dates: First submitted 2012-11-27; First posted 2012-12-04 (Estimated); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Colorectal Cancer
Keywords: Selective decontamination of the digestive tract; anastomotic leakage; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Anastomotic Leak | interventions — Colistin; Tobramycin; Amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard treatment (No Intervention): Standard treatment for colorectal cancer
- Selective decontamination of the digestive tract (SDD) (Experimental): Standard treatment + SDD perioperatively 4 times daily 10 ml of SDD suspension, consisting of 100mg colistin sulfate, 80mg tobramycin and 500mg of amphotericin B.
  SDD treatment starts 3 days before surgery and is continued until at least 3 days postoperatively.
  Interventions: Drug: Selective decontamination of the digestive tract (SDD) (colistin sulfate, tobramycin, amphotericin B)

INTERVENTIONS:
Drug: Selective decontamination of the digestive tract (SDD) (colistin sulfate, tobramycin, amphotericin B) — SDD suspension contains per dose of 10 ml 100 mg colistin sulfate, 80 mg tobramycin and 500 mg amphotericin B
  Other Names: SDD
  Arms: Selective decontamination of the digestive tract (SDD)

SUMMARY:
The primary objectives of this randomized clinical trial are to evaluate if perioperative SDD can reduce clinical anastomotic leakage rate and its septic consequences as well as other infectious complications. By reduction of septic complications long-term oncological outcome might simultaneously improve.

DETAILED DESCRIPTION:
Rationale:

Infectious complications and especially anastomotic leakage severely impede the recuperation of patients following colorectal cancer surgery. When the normal gut barrier fails such as in anastomotic leakage, pathogenic microorganisms like Gram-negative bacteria enter the circulation and may cause severe sepsis which is associated with considerable mortality. Moreover, anastomotic leakage has a negative impact on colorectal cancer prognosis. Selective decontamination of the digestive tract (SDD) is a prophylaxis regimen that employs oral nonabsorbable antibiotics to eradicate pathogenic micro-organisms like Gram-negative bacteria.

Objective:

The primary objectives of this randomized clinical trial are to evaluate if perioperative SDD can reduce clinical anastomotic leakage rate and its septic consequences as well as other infectious complications. By reduction of septic complications long-term oncological outcome might simultaneously improve. Secondary objectives are a decline in reoperation rate, in-hospital mortality, readmission rate, duration of hospital stay and ICU admission, non-infectious complications, improvement of quality of life and reduction of costs.

Study design:

A randomised multicenter clinical trial comparing perioperative SDD in addition to standard antibiotic prophylaxis with standard antibiotic prophylaxis alone in patients with colorectal cancer who undergo elective surgical resection with curative intent.

Study population:

Patients 18 years or older are eligible for inclusion when they are diagnosed with colon or rectal cancer without signs of distant metastases. Patients may be scheduled for either laparoscopic or open resection with curative intent, including construction of an anastomosis (either with or without diverting stoma). Patients are not eligible for inclusion in case of concomitant metastases or acute obstruction.

Intervention:

Patients are randomly allocated for either perioperative SDD (intervention group) including standard antibiotic prophylaxis or standard treatment (including standard antibiotic prophylaxis alone) (control group). The solution containing SDD is orally taken 4 times daily, starting 3 days before surgery and continued until normal bowel passage or at least 3 days after surgery. Both groups receive a single preoperative intravenous dose of 1000 mg Cefazoline and 500 mg Metronidazole, which is the current standard antibiotic prophylaxis.

Main study parameters/endpoints:

The main study parameter is anastomotic leakage. The research hypothesis refers to an estimated decrease in anastomotic leakage rate in the SDD treated group (from 9% to 4%). As anastomotic leakage has been shown unfavourable forlong term oncological outcome, we presume an improvement in disease free survival, which serves as important secondary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Elective colon and rectal cancer surgery with primary anastomosis
* Or elective colorectal surgery for suspected carcinoma
* No evidence of distant metastases (preoperative CT-abdomen and X-thorax or CTthorax)
* Procedure either with or without diverting stoma
* Both laparoscopic and open surgery
* Informed consent
* Aged 18 years or older

Exclusion Criteria:

* Previous colorectal malignancy
* Current malignancy which is now undergoing treatment
* Inflammatory bowel disease (Crohn's disease or ulcerative colitis)
* Previous surgery for diverticular disease
* Performance status ASA 4 or higher (American Society for Anaesthesiologists)
* Expected adverse reactions/allergies for study medication
* Prednisone use > 5 mg per day
* Familial adenomatous polyposis coli (FAP; Lynch syndrome), Hereditary Non Polyposis Colorectal Cancer (HNPCC)
* Mental disorder/unable to give informed consent
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2013-01; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
anastomotic leakage and/or abscess | 30 days postoperatively
  clinical and/or radiological evidence of anastomotic dehiscence requiring surgical or radiological (re)intervention.

SECONDARY OUTCOMES:
Disease free survival | 3 and 5 years after inclusion

OTHER OUTCOMES:
Other postoperative infectious complications | 30 days postoperatively
  pneumonia, urinary tract infections, surgical site infections, wound dehiscence, (remote) intraabdominal abscess
Non-infectious complications | 30 days postoperatively
  cardiac failure, cerebrovascular events, deep venous thrombosis
In-hospital mortality | 30 days postoperatively
Readmission rate | 5 years postoperatively
Reoperation rate | 5 years postoperatively
Duration of hospital stay | 30 days postoperatively
Quality of life (quality adjusted life years) | 2 years postoperatively
In hospital and out-of-hospital costs | 5 years postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: H.J. Bonjer, Md, PhD, FRCSC, Principal Investigator — Amsterdam UMC, location VUmc; G.S.A. Abis, MD, MSc, Study Director — Amsterdam UMC, location VUmc
Locations (5):
- Netherlands (5):
  - Slotervaart Ziekenhuis, Amsterdam
  - VU University Medical Center, Amsterdam
  - Kennemer Gasthuis, Haarlem
  - Spaarne Ziekenhuis, Hoofddorp
  - WestFries Gasthuis, Hoorn

REFERENCES:
- [Derived] Abis GSA, Stockmann HBAC, Bonjer HJ, van Veenendaal N, van Doorn-Schepens MLM, Budding AE, Wilschut JA, van Egmond M, Oosterling SJ; SELECT trial study group. Randomized clinical trial of selective decontamination of the digestive tract in elective colorectal cancer surgery (SELECT trial). Br J Surg. 2019 Mar;106(4):355-363. doi: 10.1002/bjs.11117. Epub 2019 Feb 25. PMID 30802304
- [Derived] Abis GS, Oosterling SJ, Stockmann HB, van der Bij GJ, van Egmond M, Vandenbroucke-Grauls CM, Bonjer HJ. Perioperative selective decontamination of the digestive tract and standard antibiotic prophylaxis versus standard antibiotic prophylaxis alone in elective colorectal cancer patients. Dan Med J. 2014 Apr;61(4):A4695. PMID 24814583